CLINICAL TRIAL: NCT06952335
Title: The Impact Of Respiratory Neuromuscular Stimulation On Patients With Invasive Mechanical Ventilation: A Prospective Randomized Crossover Physiological Study
Brief Title: The Impact Of Respiratory Neuromuscular Stimulation On Patients With Invasive Mechanical Ventilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Head of Emergency and Critical Care Center, Capital Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024-099-002
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-08

CONDITIONS: Mechanical Ventilation; Neuromuscular Electrical Stimulation (NMES)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phrenic nerve stimulation (PNS) at 8mA (Experimental): Phrenic nerve stimulation is applied at 8mA.
  Interventions: Procedure: Phrenic nerve stimulation at 8mA
- Phrenic nerve stimulation (PNS) at 15mA (Experimental): Phrenic nerve stimulation is applied at 15mA
  Interventions: Procedure: Phrenic nerve stimulation at 15mA
- Phrenic nerve stimulation (PNS) at 15mA combined with phrenic-abdominal stimulation at 15mA (Experimental): Phrenic nerve stimulation (PNS) at 15mA combined with phrenic-abdominal stimulation at 15mA is applied.
  Interventions: Procedure: Phrenic nerve stimulation at 15mA combined with phrenic-abdominal stimulation at 15mA

INTERVENTIONS:
Procedure: Phrenic nerve stimulation at 8mA — Phrenic nerve stimulation (PNS) at 8mA is applied.
  Arms: Phrenic nerve stimulation (PNS) at 8mA
Procedure: Phrenic nerve stimulation at 15mA — Phrenic nerve stimulation (PNS) at 15mA is applied.
  Arms: Phrenic nerve stimulation (PNS) at 15mA
Procedure: Phrenic nerve stimulation at 15mA combined with phrenic-abdominal stimulation at 15mA — Phrenic nerve stimulation (PNS) at 15mA combined with phrenic-abdominal stimulation at 15mA is applied.
  Arms: Phrenic nerve stimulation (PNS) at 15mA combined with phrenic-abdominal stimulation at 15mA

SUMMARY:
Mechanical ventilation (MV) is an important treatment measure for critically ill patients in the intensive care unit (ICU). MV is widely used in the treatment of respiratory failure and is also one of the important means of life support for critically ill patients after surgery. Although the use of MV has significantly reduced the mortality rate of critically ill patients, MV is also a double-edged sword. A large amount of evidence shows that it can lead to complications such as ventilator-induced diaphragmatic dysfunction (VIDD) . In a retrospective study, it was first found and proposed that long-term MV can lead to diaphragmatic atrophy. Later, a prospective clinical study conducted by Le Bourdelles et al. provided direct evidence to support this conjecture. Continuous use of mechanical ventilation for 48 hours can cause diaphragmatic atrophy and contractile dysfunction. Therefore, effectively preventing diaphragmatic atrophy is of great significance for the outcome of patients with mechanical ventilation.

Respiratory NMES has been used in clinical practice for decades. Previous studies have shown that electrical stimulation of a certain intensity applied to the respiratory neuromuscular can increase the excitability of the phrenic nerve, enhance diaphragmatic contraction, increase the range of diaphragmatic movement, and improve lung ventilation. In addition to the diaphragm, the abdominal muscles are also an important part of the respiratory muscles and an important supplement to the inspiratory muscles. Studies have shown that electrical stimulation of the abdominal muscles can retrain the expiratory muscles, increase muscle strength, induce expiratory muscle contraction through repeated afferent stimulation of the abdominal muscles, increase intra-abdominal pressure, facilitate the upward movement of the diaphragm, reduce thoracic pressure and lung volume, and thus improve the ability of expiration and expectoration. Electrical stimulation of the abdominal muscles has received increasing attention as a supplement to inspiratory muscle training, and many foreign literatures have reported on the improvement of respiratory function by abdominal muscle stimulation. At present, some domestic scholars have also reported that simultaneous stimulation of the phrenic nerve and abdominal muscles can improve the quality of life and prognosis of patients. However, there are few studies on how simultaneous stimulation of the diaphragm and abdominal muscles can improve the physiological effect indicators of the respiratory system, especially the impact on respiratory drive and inspiratory effort. Animal model studies have shown that electrical stimulation of the phrenic nerve in rabbits can significantly reduce the central drive of the diaphragm and the conduction function of the phrenic nerve after diaphragmatic fatigue, and the reduction of central drive may be a self-protective mechanism of the body. An observational study abroad suggested that percutaneous diaphragmatic electrical stimulation can control WOB within four-fifths of the normal range 96.8% of the time. This study is dedicated to applying respiratory NMES to study the impact on the physiological parameters of patients with invasive mechanical ventilation, providing a theoretical basis for its clinical application in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 80 years;
2. Mechanical ventilation duration > 48 hours;
3. Hemodynamically stable;
4. RASS score ranging from 1 to -2.

Exclusion Criteria:

1. Having a pacemaker implanted;
2. Unhealed surgical wounds in the chest or abdomen;
3. Pregnant women and lactating women;
4. History of recent airway surgery or trauma;
5. Surgery in the neck, chest, or upper abdomen;
6. Intracranial hypertension;
7. Contraindications for esophageal pressure catheter placement;
8. Withdrawal of life support.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Tidal swing of esophageal pressure | From enrollment to the end of treatment at 4 hours
  Tidal swing of esophageal pressure will be measured
Esophageal pressure-time product | From enrollment to the end of treatment at 4 hours
  Esophageal pressure-time product will be measured.
Inspiratory muscle pressure | From enrollment to the end of treatment at 4 hours
  Inspiratory muscle pressure will be measured.
Dynamic transpulmonary pressure | From enrollment to the end of treatment at 4 hours
  Dynamic transpulmonary pressure will be measured.

SECONDARY OUTCOMES:
Respiratory rate | From enrollment to the end of treatment at 4 hours
  Respiratory rate will be measured.
Tidal volume | From enrollment to the end of treatment at 4 hours
  Tidal volume will be measured.
Heart rate | From enrollment to the end of treatment at 4 hours
  Heart rate will be measured.
Mean blood pressure | From enrollment to the end of treatment at 4 hours
  Mean blood pressure will be measured.
Critical care pain observation tool (CPOT) scale | From enrollment to the end of treatment at 4 hours
  Critical care pain observation tool (CPOT) scale will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No